CLINICAL TRIAL: NCT06040021
Title: Integrated Analysis of Multi-center Cohorts and Bulk RNA-sequencing Data Reveal Distinct Metastatic Phenotypes Between Early-onset and Late-onset Colorectal Cancer
Brief Title: Distinct Metastatic Phenotypes Between Early-onset and Late-onset Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, Professor, Fudan University
Other Study IDs: FDU-EOCRC
Record Dates: First submitted 2023-09-11; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Early-onset Colorectal Cancer; Late-onset Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EOCRC: Patients aged<50 with colorectal cancer between 2008 and 2018 in Fudan university Shanghai cancer center.
  Interventions: Other: standardized treatment
- IOCRC: Patients aged between 50 to 70 with colorectal cancer between 2008 and 2018 in Fudan university Shanghai cancer center.
  Interventions: Other: standardized treatment
- LOCRC: Patients aged between≥70 with colorectal cancer between 2008 and 2018 in Fudan university Shanghai cancer center.
  Interventions: Other: standardized treatment

INTERVENTIONS:
Other: standardized treatment — Patients enrolled in these 2 cohorts all received standardized treatment of colorectal cancer.

SUMMARY:
The clinical and pathological features of early-onset colorectal cancer (EOCRC) differ from those of late-onset colorectal cancer (LOCRC). Our research aims to thoroughly elucidate the distinctions between them by analyzing clinical prognosis, metastatic patterns, gene expression, and genomic mutation profiles. Our deliberation will uncover latent strategies for personalized therapeutic of both EOCRC and LOCRC.

ELIGIBILITY:
Inclusion Criteria:

* The initial diagnosis of colonoscopy and pathology belongs to colorectal cancer;
* Patients should sign an informed consent form after fully understanding the purpose, procedures and potential risks of the study, indicating their voluntary participation in the research.

Exclusion Criteria:

* Patients with obvious local or systemic severe infection;
* Acute abdomen: intestinal obstruction, peritonitis, intestinal perforation;
* Have a systemic underlying disease that has not been controlled, or is unstable;
* Patients with poor physical fitness or serious other organic diseases who cannot tolerate anesthesia and surgery;
* Women during pregnancy, perinatal and lactation;
* Patients with severe mental disorders (such as schizophrenia, bipolar disorder, etc.) or patients who are mentally incapable or unable to understand the requirements for participation in the study.

Ages: 16 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with colorectal cancer hospitalized in Fudan university Shanghai cancer center.
Sampling Method: Non-Probability Sample
Enrollment: 15244 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
OS | 5 years after intervention
  overall survival